CLINICAL TRIAL: NCT01565954
Title: Systematic Evaluation of Sleep Respiratory Disorders During Sleep in Children With Sickle Cell Disease
Brief Title: Sleep Respiratory Disorders Evaluation in Sickle Cell Disease Children
Acronym: SOMMEDREP
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: P110102; 2011-005029-31 (EudraCT Number)
Record Dates: First submitted 2012-03-27; First posted 2012-03-29 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2018-02

CONDITIONS: Sickle Cell Disease; Respiration Disorders
Keywords: Sickle Cell Disease; Respiration Disorders; Polysomnography
MeSH Terms: conditions — Anemia, Sickle Cell; Respiration Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
In Sickle cell disease children, sleep respiratory abnormalities are risk factors for vaso-occlusive complications, as well as cerebral vasculopathy.

A 18 months follow-up children with sickle cell disease evaluating sleep respiratory problems frequency and etiology, as well as their influence on sickle cell disease complications.

DETAILED DESCRIPTION:
* Inclusion visit with physical examination. A 2.9 ml blood sample will be necessary, if not done within the framework of care within 6 months for: CBC (Cell Blood Count), reticulocytes counts (1.2 ml of blood), liver enzymes, electrolytes, urea, creatininemia (1,2 ml of blood) and fetal hemoglobin (0.5 ml of blood). - A complete standardized examination including nasopharynx endoscopy, if not yet done in usual care, to identified upper airway obstruction
* A standardized pneumology evaluation to identified obstructive lung symptomatology
* An ambulatory polysomnography will be performed within days following inclusion, during sleep and will allow electroencephalogram recording, oculomotricity, muscles (mentalis muscles and tibialis anterior) movements, electrocardiogram and respiratory activity recording.

The steering committee will classify the children in three populations based on their exam results:

* Group 1: no abnormality in polysomnography
* Group 2: obstructive sleep-related disorder
* Group 3: isolated sleep hypoxemia for group3, patients will have a new ambulatory polysomnography.

ELIGIBILITY:
Inclusion Criteria:

* Sickle cell disease children with either sickle cell anemia, compound heterozygozity SB0-thalassemia, or SDPunjab,
* no prior transfusion program within 3 months,
* no prior treatment with hydroxycarbamide within 3 months,
* Aged 2 to 6 years,
* Parents or tutors signed informed consent,
* Prior physical examination,
* Social security insurance.

Exclusion criteria:

* Encephalopathy
* Other disease that could interfere with protocol exams realization
* Nitrous oxide analgesia contre-indication
* Conventional hospitalization in the past 3 weeks

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The objective of this study is to provide an early curative treatment for homozygous sickle cell children in age group of 2 to 6 years based on the anomalies identified in polysomnography. The choice of the age of 2 to 6 is linked to the peak risk of onset of cerebrovascular occlusive complications in this age
Sampling Method: Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Vaso-occlusive and cerebral complications frequency | 18 months
  Vaso-occlusive complications frequency and abnormal transcranial doppler (TCD) during the 18 months of follow up (cohort study) 3 subpopulations will be identified upon polysomnographic results:
  * Group 1: normal polysomnography
  * Group 2: sleep abnormalities related to obstructive upper airway disease or bronchial disease
  * Group 3: sleep abnormalities associated with non-obstructive pattern and isolated hypoxemia identified. The therapeutic trial will be done on this group.

SECONDARY OUTCOMES:
Respiratory sleep abnormalities frequency | 18 months
  Respiratory sleep abnormalities frequency in a population of young sickle cell disease children.
Relationship between sleep abnormalities and transcranial doppler abnormalities | 2 months
  Analyze the relationship between sleep respiratory and non-respiratory abnormalities and transcranial doppler abnormalities
Polysomnography relevance compared to sleep ventilatory polygraphy | 2 months
  Polysomnography relevance compared to sleep ventilatory polygraphy in diagnosis of sleep abnormalities

CONTACTS AND LOCATIONS:
Overall Officials: Malika BENKERROU, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Assistance Publique - Hôpitaux de Paris, Paris, France